CLINICAL TRIAL: NCT06623058
Title: Accupower ® HCV Performance Evaluation Quant Kit Bioneer Existation™FA 96/384
Acronym: BIOPERF-HCV
Status: Not yet recruiting | Type: Observational
Sponsor: CerbaXpert (Other)
Collaborators: Bioneer Corporation (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2024-A01285-42; 2024-A01285-42 (Other: ANSM)
Record Dates: First submitted 2024-09-30; First posted 2024-10-02 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-09

CONDITIONS: HEPATITIS C (HCV)
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood sample frome hepatitis C infected patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Infected patients with hepatitis C virus: Infected patients with hepatitis C virus

SUMMARY:
As part of the CE marking of a hepatitis C diagnostic kit, the South Korean manufacturer Bioneer wishes to set up a performance study in France in accordance with the IVDR (RE 2017/746).

Cerba Xpert CRO of the Cerba Healthcare group promoted this performance study by setting up a prospective collection of blood samples from patients suffering from the virus hepatitis C and whose viral load is positive. This prospective collection will be carried out in 4 laboratories of the Cerba Healthcare group.

DETAILED DESCRIPTION:
Viral hepatitis are primarily human systemic infections caused by viruses hepatic diseases which cause damage to the liver by hepatocyte infection of the virus and/or a host immune response to the virus. (1) Hepatitis is grouped into five types (A, B, C, D, E) and is mainly transmitted by parenteral, sexual and fetomaternal.(2) The hepatitis C virus (HCV) was discovered in 1989.(3) It is an RNA virus that belongs to the family Flaviviridae.(4) Infection with the hepatitis C virus is characterized by clinical signs such as such as jaundice, asthenia, anorexia. In approximately 30% (15% to 45%) of infected people, the virus is spontaneously eliminated within six months following infection, without any treatment. (5) For the remaining 70% (55% to 85%), the infection will progress to a chronic form. In patients chronic, the risk of cirrhosis is 15% to 30% in the 20 years following infection. (5) A assessment of liver damage and virus replication in the blood is made before starting treatment.(6) Detection/quantification of HCV RNA in serum or plasma must therefore be available before to initiate antiviral treatment. HCV RNA must be tested for by a sensitive test giving a result viral load expressed in IU/ml and Log IU/ml. (6) Monitoring of response to treatments is done also by the detection of viral RNA, particularly at 12 weeks post-treatment where a viral load undetectable is a sign of effective treatment and healing. (6) On the European market, quantitative determination of hepatitis C viral load as part of Diagnosis and monitoring of the disease is done by real-time PCR which is the reference technique.(7) As part of routine care, there are several diagnostic PCR kits that can be used on plasma or serum. Today, there are no CE approved PCR kits that allow the quantification of viral RNA at the both serum and plasma. Our study will make it possible to evaluate the performance of the Bionner kit PCR kit ACCUPOWER Quant Kit Bioneer Existation™FA 96/384 on serum and plasma of affected patients hepatitis C.

ELIGIBILITY:
Inclusion Criteria:

The patient to be included in this study must be able to understand the purpose of the research, in order to to give free and informed consent.

* Subject aged over 18
* Subject presenting at the investigation center and meeting one of these two criteria:

  * Subject presenting with a prescription for HCV viral load determination
  * Subject whose HCV infection is previously confirmed by CE marked tests.
* Subject capable of understanding the purpose of the research having given express free and informed consent
* Subject affiliated to or beneficiary of a social security system

Exclusion Criteria:

Protected subject: adult under guardianship, curatorship or other legal protection, deprived of liberty by judicial decision or administrative Subject participating in a clinical study/receiving investigational treatment

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Infected patients with hepatitis C virus
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
Commutability between serum and plasma hepatitis C viral load results with the ACCUPOWER HCV Quant Kit Bioneer Existation™FA 96/384. | 4 months
  The submitted protocol is carried out as part of a 'commutability' study, that is to say for Compare two matrix types on the Accupower ® HCV Quant Kit Bioneer Existence™FA 96/384. Indeed, for these two matrices to be claimed in the IFU of the kit it is necessary to prove that the two matrices give the same result.
  The planned size of the evaluable cohort is 45 patients included over a period of 4 month. This size is justified by the recommendations of the applicable CLSI EP09 guide.
  This guide details the use of several mathematical models that guarantee robust analysis even on a small cohort size. The operating methodology of the results is detailed below, taken from the recommendations of the CLSI EP09 guide

CONTACTS AND LOCATIONS:
Locations (1):
- Cerba Xpert, Frépillon, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No